CLINICAL TRIAL: NCT01613079
Title: Evaluation of Oral T2 (Chloroform/Methanol Extract of Tripterygium Wilfordii Hook F) in the Treatment of RA Patients With Clinical Efficacy and Safety.
Brief Title: Efficacy and Safety of Tripterygium Wilfordii in Patients With Rheumatoid Arthritis
Acronym: TRIFRA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xuan Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIFRA
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Methotrexate; Tripterygium
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methotrexate (Placebo Comparator): Patients were treated with methotrexate alone.
  Interventions: Drug: Methotrexate
- T2 (Experimental): Patients were treated with oral T2 (chloroform/methanol extract of Tripterygium wilfordii Hook F).
  Interventions: Drug: Tripterygium wilfordii Hook F
- MTX+T2 (Experimental): The patients were treated with methotrexate and T2.
  Interventions: Drug: Tripterygium wilfordii Hook F; Drug: Methotrexate

INTERVENTIONS:
Drug: Tripterygium wilfordii Hook F — Oral T2(Tripterygium wilfordii Hook F) 20mg thrice daily for 24 weeks.
  Arms: MTX+T2; T2
Drug: Methotrexate — Oral methotrexate 7.5-12.5mg per week for 24 weeks. The starting dose was 7.5mg per week, then increased to 12.5mg（max 0.3mg/Kg） per week in 4 weeks. Folic acid at the dose of 10mg per week were applied to all patients.
  Arms: MTX+T2; Methotrexate

SUMMARY:
Evaluation of oral T2 (chloroform/methanol extract of Tripterygium wilfordii Hook F) in the treatment of RA patients with clinical efficacy and safety.Open-labeled, randomized, prospective multi-center clinical trial. Observation period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with informed consent
* Diagnosed with rheumatoid arthritis as determined by meeting the 2010 ACR/EULAR classification criteria and has had rheumatoid arthritis for at least 6 weeks
* Swollen joint (SJC)≥3 and tender joint count(TJC)≥5
* ESR >28 mm/hr or C-reactive protein > 20 mg/L

Exclusion Criteria:

* Pregnant, lactating or further fertility requirements
* Previous treated with methotrexate or biologic DMARD.
* Active or chronic infection, including HIV, HCV, HBV, tuberculosis
* Patient with cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
ACR50 | 24 weeks.
  The proportion of patients achieving ACR50.

SECONDARY OUTCOMES:
Radiology outcome | 24 weeks
  The change in X-Ray from baseline to week 24.
DAS28 | 24 weeks
  The change in DAS score from baseline to week 24.
ACR20/70 | 24 weeks
  The proportion of patients achieving ACR20 & ACR70.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou YZ, Zhao LD, Chen H, Zhang Y, Wang DF, Huang LF, Lv QW, Liu B, Li Z, Wei W, Li H, Liao X, Liu H, Liu X, Jin H, Wang J, Fei YY, Wu QJ, Zhang W, Shi Q, Zheng WJ, Zhang FC, Tang FL, Lipsky PE, Zhang X. Comparison of the impact of Tripterygium wilfordii Hook F and Methotrexate treatment on radiological progression in active rheumatoid arthritis: 2-year follow up of a randomized, non-blinded, controlled study. Arthritis Res Ther. 2018 Apr 10;20(1):70. doi: 10.1186/s13075-018-1563-6. PMID 29636089
- [Derived] Lv QW, Zhang W, Shi Q, Zheng WJ, Li X, Chen H, Wu QJ, Jiang WL, Li HB, Gong L, Wei W, Liu H, Liu AJ, Jin HT, Wang JX, Liu XM, Li ZB, Liu B, Shen M, Wang Q, Wu XN, Liang D, Yin YF, Fei YY, Su JM, Zhao LD, Jiang Y, Li J, Tang FL, Zhang FC, Lipsky PE, Zhang X. Comparison of Tripterygium wilfordii Hook F with methotrexate in the treatment of active rheumatoid arthritis (TRIFRA): a randomised, controlled clinical trial. Ann Rheum Dis. 2015 Jun;74(6):1078-86. doi: 10.1136/annrheumdis-2013-204807. Epub 2014 Apr 14. PMID 24733191